CLINICAL TRIAL: NCT04903912
Title: Campania Registry On Peripheral Artery Disease
Acronym: CARE-PAD
Status: Recruiting | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Giuseppe Giugliano, Professor, Federico II University
Other Study IDs: 95/21
Record Dates: First submitted 2021-04-21; First posted 2021-05-27 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Peripheral Artery Disease
Keywords: Outcome; Peripheral revascularization
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Clinical Laboratory Techniques

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Vascular ultrasound or other imaging methods according to current guidelines — Peripheral vascular ultrasound / ankle/brachial index / CT angiography / MR angiography / angiography
Diagnostic Test: Laboratory tests — Metabolic profile and platelet reactivity
Drug: Medical treatment according to current guidelines — Antithrombotic drugs, lipid-lowering drugs, antihypertensive drugs, and pharmacotherapy to increase walking capacity according to current guidelines
Procedure: Endovascular od surgical peripheral revascularizations — Endovascular od surgical peripheral revascularizations according to current guidelines

SUMMARY:
The CAmpania REgistry on Peripheral Artery Disease (CARE-PAD) is a single-center observational study which has the purpose to collect clinical, laboratory, instrumental, procedural and follow-up data and to evaluate the outcome of peripheral artery disease (PAD) patients.

DETAILED DESCRIPTION:
PAD patients had widespread atherosclerosis and show a worse prognosis than patients with coronary artery disease alone. The CAmpania REgistry on Peripheral Artery Disease (CARE-PAD) is a single center observational study conducted at the Department of Advanced Biomedical Sciences of the Federico II University of Naples which aims to collect clinical, laboratory, instrumental, procedural and follow-up data and to evaluate short, medium and long term outcome of PAD patients. Patients with established diagnosis of peripheral arterial disease according to current international guidelines will be included in the observational study. The overall duration of the study will be 10 years. The presence of PAD will be confirmed based on clinical and instrumental criteria:

* Intermittent claudication and/or critical limb ischemia with presence of haemodynamically significant stenosis/occlusion of the lower limb arteries detected by ultrasound and/or other imaging methods or with ankle/brachial index (ABI) ≤ 0.90.
* Carotid stenosis of at least 50% at ultrasound and/or at other imaging methods
* Abdominal aortic aneurysm (≥3 cm) found at ultrasound and/or other imaging methods.
* History of peripheral/carotid revascularization or of aortic aneurysm treatment.

All patients will be managed according to current guidelines and will receive maximal antiatherosclerotic medical therapy to improve cardiovascular prognosis and, if clinically indicated, could undergo peripheral revascularization procedures to improve symptoms and/or limb prognosis. The choice of the revascularization procedure will be based on careful individual evaluation and will take into account, in accordance with current guidelines, several variables such as clinical characteristics, comorbidities, individual surgical risk and feasibility of the percutaneous peripheral revascularization procedure.

ELIGIBILITY:
Inclusion Criteria:

Confirmed diagnosis of peripheral artery disease as follows (one or more of the following):

* Intermittent claudication with presence of hemodynamically significant stenosis/occlusion of lower limb arteries or pathological ABI (≤ 0.90);
* Critical limb ischemia with presence of hemodynamically significant stenosis/occlusion of lower limb arteries or pathological ABI (≤ 0.90);
* Presence of carotid stenosis of at least 50%;
* Presence abdominal aortic aneurysm (≥ 3 cm);
* History of peripheral/carotid revascularization or of aortic aneurysm treatment.

Exclusion Criteria:

Refusal to sign the informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected di peripheral artery disease
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2031-05-01 (Estimated); Study Completion 2031-05-01 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiovascular Events (MACE) | 10 years
  Death from cardiovascular causes Non-fatal myocardial infarction Non-fatal stroke Ruptured aortic aneurysm
Major Adverse Limb Events (MALE) | 10 years
  Development of critical limb ischemia Peripheral revascularization for development of severe ischemia Any amputation

SECONDARY OUTCOMES:
Any adverse event other than MACE or MALE | 10 years
  Any-cause death or any adverse cardiovascular event other than MACE or MALE (transient ischemic attack, unstable angina, any coronary, carotid or peripheral revascularization);
Bleeding events | 10 years
  Periodic assessment of bleeding events according to the BARC classification
Instrumental assessment of functional capacity | 10 years
  Instrumental assessment of maximum walking distance (MWD) (meters)
Assessment of quality of life | 10 years
  Quality of life will be periodically assessed by evaluating change in EuroQol (EQ) - 5 Dimensions (5D) - 5 Levels (5L) questionnaire (EQ-5D-5L™) from baseline (range 0-1 with 0 expressing the worst health state and 1 the best)
Assessment of functional status | 10 years
  Walking capacity will be periodically assessed by evaluating change in Walking Impairment Questionnaire (WIQ) from baseline; range 0-100%, where 0% represents the lowest possible score (ie, answering "unable" for all questions in that category) and 100% represents the highest possible score (ie, indicating "none" with regard to difficulty for all questions in that category)
Assessment of frailty in geriatric population | 10 years
  All patients aged 65 and over will be assessed for frailty through the Multidimensional Prognostic Index (MPI), a multidimensional score (range 0-1; 0.00-0.33 mild frailty; 0.34-0.66 moderate frailty; 0.67-1.00 severe frailty).
Assessment of functional status in geriatric population | 10 years
  Functional status for all patients aged 65 and over will be further assessed with Short Physical Performance Battery (SPPB) (pathologic if ≤ 8 in males and ≤ 7 in females) and Handgrip strength (pathologic in men for ≤ 29 kg when BMI ≤ 24 kg/m2 or ≤ 30 kg when BMI 24,1-28 kg/m2 or ≤ 32 kg when BMI > 28 kg/m2; pathologic in women for ≤ 17 kg when BMI ≤ 23 kg/m2 or ≤ 17,3 kg when BMI 23,1-26 kg/m2 or ≤ 18 kg when BMI 26,1-29 kg/m2 or ≤ 21 kg when BMI > 29 kg/m2)
Assessment of cognitive performance in geriatric population | 10 years
  Cognitive status for all patients aged 65 and over will be assessed with: Mini Mental State Examination (MMSE) (< 24/30 normal; 18-24/30 mild cognitive impairment; 12-18/30 moderate cognitive impairment; <12/30 severe cognitive impairment); Clock Drawing Test (pathologic if ≤ 3/5); Digit span forward (pathologic if ≤ 4/16; borderline if 4-5/16; normal if > 5/16) and backward (pathologic if ≤ 3/16; borderline if 3-4/16; normal if > 4/16); Trail making test A (pathologic if > 78 seconds) and B (pathologic if > 273 seconds); Hospital Anxiety and Depression Scale (HADS) ( 0-7 normal; 8-10 borderline; 11-21 pathologic)
Evaluation of lipid profile | 10 years
  Periodic evaluation of lipid profile (total cholesterol, LDL cholesterol, HDL cholesterol, triglycerides in mg/dl)
Evaluation of metabolic profile | 10 years
  Periodic evaluation of glucose levels (mg/dl)
Atherosclerosis progression | 10 years
  Periodical ultrasound evaluation of the progression of atherosclerosis at different vascular districts [measurement of degree of stenosis (%)]
P2Y12 Reaction Unit (PRU) at VerifyNow | 28 days
  Platelet aggregation assessed with VerifyNow ADP test in patients who start dual antiplatelet therapy or dual antithrombotic therapy
Area under the curve (AUC) at Multiplate with ADP test | 28 days
  Platelet aggregation assessed with Multiplate ADP test in patients who start dual antiplatelet therapy or dual antithrombotic therapy
Inhibition of platelet activity (IPA, %) with LTA-ADP 20 µmol/l | 28 days
  Platelet inhibition assessed with LTA-ADP 20 µmol/l in patients who start dual antiplatelet therapy or dual antithrombotic therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Advanced Biomedical Sciences, University of Naples "Federico II", Naples, Italy

REFERENCES:
- [Background] Aboyans V, Ricco JB, Bartelink MEL, Bjorck M, Brodmann M, Cohnert T, Collet JP, Czerny M, De Carlo M, Debus S, Espinola-Klein C, Kahan T, Kownator S, Mazzolai L, Naylor AR, Roffi M, Rother J, Sprynger M, Tendera M, Tepe G, Venermo M, Vlachopoulos C, Desormais I; ESC Scientific Document Group. 2017 ESC Guidelines on the Diagnosis and Treatment of Peripheral Arterial Diseases, in collaboration with the European Society for Vascular Surgery (ESVS): Document covering atherosclerotic disease of extracranial carotid and vertebral, mesenteric, renal, upper and lower extremity arteriesEndorsed by: the European Stroke Organization (ESO)The Task Force for the Diagnosis and Treatment of Peripheral Arterial Diseases of the European Society of Cardiology (ESC) and of the European Society for Vascular Surgery (ESVS). Eur Heart J. 2018 Mar 1;39(9):763-816. doi: 10.1093/eurheartj/ehx095. No abstract available. PMID 28886620
- [Background] Erbel R, Aboyans V, Boileau C, Bossone E, Bartolomeo RD, Eggebrecht H, Evangelista A, Falk V, Frank H, Gaemperli O, Grabenwoger M, Haverich A, Iung B, Manolis AJ, Meijboom F, Nienaber CA, Roffi M, Rousseau H, Sechtem U, Sirnes PA, Allmen RS, Vrints CJ; ESC Committee for Practice Guidelines. 2014 ESC Guidelines on the diagnosis and treatment of aortic diseases: Document covering acute and chronic aortic diseases of the thoracic and abdominal aorta of the adult. The Task Force for the Diagnosis and Treatment of Aortic Diseases of the European Society of Cardiology (ESC). Eur Heart J. 2014 Nov 1;35(41):2873-926. doi: 10.1093/eurheartj/ehu281. Epub 2014 Aug 29. No abstract available. PMID 25173340
- [Background] Fowkes FG, Rudan D, Rudan I, Aboyans V, Denenberg JO, McDermott MM, Norman PE, Sampson UK, Williams LJ, Mensah GA, Criqui MH. Comparison of global estimates of prevalence and risk factors for peripheral artery disease in 2000 and 2010: a systematic review and analysis. Lancet. 2013 Oct 19;382(9901):1329-40. doi: 10.1016/S0140-6736(13)61249-0. Epub 2013 Aug 1. PMID 23915883